CLINICAL TRIAL: NCT04654975
Title: Risk Factors and Treatment Options for Metachronic Brain Metastases After Esophagectomy for Esophageal Cancer: a Multicentric Retrospective Cohort Study (METABREC)
Brief Title: Metachronic Brain Metastases After Esophagectomy for Esophageal Cancer (METABREC)
Acronym: METABREC
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S64060
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Neoplasms; Esophagectomy; Brain Metastases
MeSH Terms: conditions — Esophageal Neoplasms; Brain Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Esophagectomy for esophageal cancer — Surgical removal of (a part of) the esophagus and surgical reconstruction with another organ (mostly stomach, but may be colon or small bowel as well)

SUMMARY:
Esophagectomy is the cornerstone of the curative treatment of esophageal carcinoma. Despite this treatment, patients can suffer from locoregional or distant metastatic disease and only a very selected group of patients can be cured: mostly those with recurrence in one single organ.

Brain metastases are rare after esophagectomy for cancer, but they have a serious impact on survival. Agressive treatment is often moren difficult for brain metastases compared to other metastases and some risk factors have been identified earlier.

There is an impression that the incidence of brain metastases in esophageal cancer patients has increased since the introduction of neoadjuvant treatment schemes. However, this is not clear yet. A potential explanation could be that chemotherapy disturbs the blood-brain-barrier, hereby facilitating the migration of tumor cells to the brain.

The purpose of this study is to retrospectively analyze the incidence and potential risk factors of brain metastases in patients who underwent esophagectomy for esophageal cancer. Patients treated between 2000 and 2019 will be included and outcome parameters are Odds Ratio for brain metastases (comparison between primary surgery and neoadjuvant treatment followed by surgery), time to recurrence and risk factors, number and characteristics of the brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving surgical treatment for esophageal cancer between 1 januari 2000 and 31 december 2019
* All types of neoadjuvant treatment followed by surgery, primary surgery or salvage surgery.
* Adenocarcinoma or squamous cell carcinoma histology

Exclusion Criteria:

* other histology type than adenocarcinoma or squamous cell carcinoma
* Hypopharyngeal carcinoma extending to the esophagus (requiring total laryngo-pharyngo-esophagectomy)
* Early esophageal carcinoma (cT IS-1a N0 M0)
* palliative esophagectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving surgical treatment for esophageal cancer between 1 januari 2000 and 31 december 2019
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Odds ratio (OR) for brain metastasis | 1 January 2000 - 1 March 2020
  Odds ratio (OR) for brain metastasis compared between primary surgery and neoadjuvant treatment plus surgery, OR for different neoadjuvant treatment regimes, corrected for gender and tumor factors (histology, stage, tumor differentiation,…) .

SECONDARY OUTCOMES:
Overall survival | 1 January 2000 - 1 March 2020
  Overall survival after diagnosis of brain metastases stratified for treatment regimens applied.
Time to recurrence | 1 January 2000 - 1 March 2020
  Time to recurrence, between incidence date of esophageal cancer and diagnosis of brainM+
Risk factors for single site brain metastasis | 1 January 2000 - 1 March 2020
  such as different neoadjuvant treatment regimes, age, gender,and tumor factors (histology, stage, tumor differentiation,…)
Number of brain metastases | 1 January 2000 - 1 March 2020
  Number of brain metastases
Characteristics of brain metastases | 1 January 2000 - 1 March 2020
  solitary/multiple; location /side in the brain; treatment) and the effects on 'OS after recurrence' (e.g. is there a significant survival benefit in patients with brainM+ if they are treated with brain-surgery and/or stereotactic radiotherapy compared to non-treated BrainM+ or palliative treatments of brainM+

CONTACTS AND LOCATIONS:
Overall Officials: Lieven P Depypere, PhD, Principal Investigator — UZ Leuven
Locations (8):
- MD Anderson Cancer Center, Houston, Texas, United States
- Universitair ziekenhuis Gent, Ghent, Belgium
- Centre Hospitalier régional Universitaire de Lille, Lille, France
- Saint James Hospital, Dublin, Ireland
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - Zuyderland MC, Heerlen
  - Erasmus MC, Rotterdam
- Karolinska Institutet, Stockholm, Sweden